CLINICAL TRIAL: NCT01424761
Title: Coenzyme Q10 in Relation to the Antioxidative Vitamins, Oxidative Stress and Inflammation in Coronary Artery Disease Patients During Statin Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: S10241
Record Dates: First submitted 2011-08-24; First posted 2011-08-29 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Experimental): Placebo:starch
  Interventions: Other: Placebo
- Coenzyme Q10 (Experimental)
  Interventions: Dietary Supplement: Coenzyme Q10

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 — Coenzyme Q10 300 mg/d (150 mg/bid)
  Other Names: Ubquionine
  Arms: Coenzyme Q10
Other: Placebo — Placebo :starch
  Arms: Placebo

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of Taiwan. American Heart Association (AHA) indicated that CVD patients with Statin therapy would decrease the recurrence of CVD. The goal for lipid lowering in CVD patients was set at the level of low-density lipoprotein cholesterol (LDL-C) below 100 mg/dL. Coenzyme Q10 is recognized as a lipid soluble antioxidant, Statin treatment might affect the level of coenzyme Q10. Therefore, the purposes of this study are going to investigate the relation of coenzyme Q10 with other antioxidant vitamins (Vitamin A and E), the markers of lipid peroxidation, antioxidant enzymes activities, and the inflammatory markers in coronary artery disease (CAD) patients during Statin therapy. The study is going to design a placebo-controlled study. The investigators will recruit coronary artery disease (CAD) patients who are identified by cardiac catheterization as having at least 50% stenosis of one major coronary artery, and healthy subjects. CAD subjects are randomly assign to placebo and coenzyme Q10 supplements (150 mg/bid = 300 mg/d) groups. Intervention is going to administration for three months. Fasting blood will be obtained in each month and determine the concentration of antioxidant vitamins, lipid peroxidation markers, antioxidant enzymes activities after intervention. Meanwhile, the investigators will measure the level of inflammatory markers in all subjects of this study. Hopefully, the results of this study could provide information of coenzyme Q10 supplementation for clinical dietitian in advising CAD patients who are under Statin therapy.

ELIGIBILITY:
Inclusion Criteria:

CAD patients is identified by cardiac catheterization as having at least 50% stenosis of one major coronary artery and under statin therapy.

Exclusion Criteria:

* age < 18 years old
* pregnancy women
* taking antioxidant vitamins supplements

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Antioxidant and inflammation | 12 weeks
  The study are going to measure the concentrations of coenzyme Q10, vitamin A and E, lipid peroxidation markers (TBARS) and antioxidant enzymes activities (catalase, glutathione peroxidase and superoxide dismutase), and the level of inflammatory markers (hs-CRP, TNF-alfa, IL-6 and adiponectin) in all subjects of this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Verterans General Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Lee BJ, Tseng YF, Yen CH, Lin PT. Effects of coenzyme Q10 supplementation (300 mg/day) on antioxidation and anti-inflammation in coronary artery disease patients during statins therapy: a randomized, placebo-controlled trial. Nutr J. 2013 Nov 6;12(1):142. doi: 10.1186/1475-2891-12-142. PMID 24192015